CLINICAL TRIAL: NCT05347823
Title: Study of Adherence to Antihypertensive Drugs and Statins in the Population of Subjects With Hypertension Followed at SIIA Centers, Using an Innovative Monitoring Based on Hair Analysis
Brief Title: Study of Adherence to Antihypertensive Drugs and Statins by Hair Analysis
Acronym: INNOVA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Collaborators: Societa Italiana dell'Ipertensione Arteriosa (Other)
Responsible Party: Sponsor
Other Study IDs: 3421CESC
Record Dates: First submitted 2022-04-21; First posted 2022-04-26 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Arterial Hypertension; Dyslipidemias; Antihypertensive Drugs; Statins; Treatment Adherence
MeSH Terms: conditions — Hypertension; Dyslipidemias; Treatment Adherence and Compliance | interventions — Hair Analysis; Blood Pressure Monitoring, Ambulatory; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples, hair samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Hair analysis for drug concentration — Sample collection for the determination of treatment adherence
  Other Names: Blood pressure monitoring; Blood sampling

SUMMARY:
The problem of adherence to long-term therapies has been known for years and occurs substantially in all countries, although with greater severity in developing countries. The investigators designed a prospective open study in which 200 patients followed for hypertension at the centers of the Italian Society of Hypertension (SIIA) adhering to the project will be evaluated on the basis of their clinical characteristics, the presence of comorbidities and the therapeutic scheme in place and will be subjected to hair sampling for the analysis of drugs of interest and their possible metabolites in this matrix. The use of the prescribed drugs is recorded along with the relevant clinical parameters and preliminarily evaluated by application of a questionnaire. At the first visit, patients who have been prescribed continuously in the 3 months preceding the study the same active ingredients will be invited to participate in the study, which involves a hair sampling. They will then be prescribed the same active ingredients according to the same scheme if the blood pressure values are within the recommended limits. When more than one antihypertensive drug is present in the therapeutic scheme, they will be prescribed in a single pill, as recommended. For patients with uncontrolled blood pressure, the therapeutic scheme will be modified with the inclusion of other active ingredients and using drug combinations when possible. Patients treated with statins will continue the treatment according to clinical indication using associations with antihypertensive drugs. Patients will be examined and re-tested 3-4 months after the first visit. The use of prescribed medications will be recorded along with clinical parameters of interest and preliminarily evaluated by application of questionnaires. At each of the two visits, the investigating physician will measure blood pressure using a semi-automatic device The 24-hour blood pressure monitoring will be used. Hair extraction ad UHPLC-QQQ/MS analysis will be performed. Concentrations of active ingredient and any metabolites in the keratin matrix are expressed in ng or fractions of ng/mg.

DETAILED DESCRIPTION:
The problem of adherence to long-term therapies has been known for years and occurs substantially in all countries, although with greater severity in developing countries.There is a positive correlation between poor adherence and mortality, as demonstrated by Simpson et al. with their analysis of data from 46,847 patients: the risk of mortality is halved for patients who take their medications appropriately compared to non-adherent patients (Simpson, 2016). It is reasonable to assume that medication non-adherence will increase as life expectancy increases, resulting in more chronic conditions to be treated.

The main areas in which monitoring adherence to therapy can play a crucial role, according to the aforementioned World Health Organization (WHO) document include primarily cardiovascular disease, The data on the use of drugs in the Italian population show dramatically low adherence to the prescribed therapy, with data of persistence in therapy at one year of 53% for antihypertensive drugs and 47% for lipid lowering drugs (OSMED). There is urgent need to promote cognitive investigations on the causes of abandonment of therapy and to have appropriate tools to assess the real adherence to therapy in the individual patient.

These two objectives can be pursued through longitudinal studies: retrospective studies related to patients for whom there is data collection and prospective studies in which the relationship between the treatment schedule, clinical characteristics of patients and medical intervention can be subjected to experimental verification. For these studies it is necessary to use analysis tools suitable to evaluate, over time, the real exposure of patients to the drugs prescribed. The analysis of pharmaceuticals (and their metabolites) in keratinized tissues, such as hair, appears to meet many needs for retrospective analytical investigation. The known and relatively constant speed of hair growth, considering that the xenobiotics incorporated at the root level remain virtually unmodified for a long time, allows to chronologically place the intake of substances in relation to their distribution along the hair shaft (see: Guidelines for Testing Drugs under International Control in Hair Sweat and Oral Fluid, UNODC, Vienna, 2014). The present investigation is a prospective open study in which 200 patients followed for hypertension at the centres of the Italian Society of Hypertension (SIIA) willing to take part will be evaluated on the basis of their clinical characteristics, the presence of comorbidities and their therapeutic scheme will be subjected to hair sampling for the analysis of drugs of interest and their possible metabolites in this matrix. The use of the prescribed drugs will be recorded along with the relevant clinical parameters and preliminarily evaluated by application of a questionnaire. At the first visit, patients who have been prescribed continuously in the 3 months preceding the study the same active ingredients will be invited to participate in the study, which involves a hair sample (about 100 mg cut from the skin, recommended length 3 cm). They will then be prescribed the same drugs according to the same scheme if the blood pressure values are within the recommended limits. When more than one antihypertensive drug is present in the therapeutic scheme, they will be prescribed as a single pill, as recommended (Hypertension Guidelines 2018, Primary Prevention 2021). For patients with uncontrolled blood pressure, the therapeutic scheme will be modified with the inclusion of other drugs and using pills with drug combinations when possible. Patients treated with statins will continue the treatment according to clinical indication using, when possible,pills containing associations with antihypertensive drugs. The same procedure will apply in case a statin is included in the therapy for clinical indication. Patients will be given two questionnaires: BMQ (Brief Medication Questionnaire); MUAH (Maastricht Utrecht Adherence in Hypertension questionnaire); MMAS (Morisky Medication Adherence Scale). This will allow a comparison of the data obtained from the questionnaires with the analytical data from the hair analysis.Patients will be examined and re-tested 3-4 months after the first visit. The use of prescribed medications will be recorded along with clinical parameters of interest and preliminarily evaluated by application of questionnaires.

At each of the two visits, the investigating physician will measure blood pressure (average of 3 measurements) at the first and second visit, using a semi-automatic device according to the European Society of Hypertension guidelines (ESH-ESC guidelines 2018): in the sitting position (measured at both arms at the first visit) and orthostatic position (3 measurements after 1 and 3 minutes) and heart rate. Ambulatory blood pressure monitoring (24-hour) will be performed within a short time interval from the first visit and the second visit.Total cholesterol, LDL and HDL cholesterol, triglyceridemia, glycemia, uricemia, creatinine, sodium, potassium, and complete blood cells count, recently performed by the patient according to clinical indications, will also be recorded.

The investigating physician will be able to acquire information about the patient, through information requested directly from the family doctor as per clinical practice.

Data management and procedures to ensure data confidentiality: Patients data will remain protected in compliance with European Union data protection regulations (EU General Data Protection Regulation 679/2016).

The collected data will be anonymized by assigning an identification code for each patient that will be reported in the data collection form. The attribution of the code and the link to the patient's name will be in an electronic card whose access is limited only to investigators at the site with protected access. To minimize the risk of unauthorized access, the hardware in which patient data will be recorded will be placed in a restricted access area accessible only to authorized personnel who need to retrieve information for professional purposes. The electronic database will be protected through the use of a username and password that will be changed periodically.

The samples will be stored for 15 years at the Institute of Forensic Medicine of the University of Verona.

The data obtained will be owned by the investigators and co-experimenters (including recruitment centers).

Analytical Methods: Hair extraction ad ultra high performance liquid chromatography (UHPLC)- triple quadrupole mass spectrometry (QQQ/MS) analysis will be performed in Verona (Prof. Franco Tagliaro, Department of Forensic Medicine). Mode of expression of results: concentrations of active ingredient and any metabolites in the keratin matrix are expressed in ng or fractions of ng/mg.

Sample size calculation: The proposed study is aimed at defining the feasibility and the necessary sample size - thus defining the objectives of an intervention study aimed at achieving a high degree of adherence to drug therapy and, consequently, to have an impact on clinical events in the population actively followed compared to the historical data and the reference population. Since this is a pilot study has not been performed an a priori calculation of sample size, but it is expected to enroll about 200 subjects in 6 months of enrollment.

Study duration: Patient Enrollment Duration: 6 months Patient Involvement: 3 months Total Study Duration: 12 months Data analysis: Data will be collected anonymously using a progressive code that can also identify the different centers. Continuous variables will be summarized through mean and standard deviation if normally distributed, and through median and interquartile range if asymmetrically distributed, while for categorical variables absolute or relative frequencies will be used. Significance of differences will be assessed by Student's t test (or the Mann-Whitney test for nonparametric analyses) for quantitative variables and by Fisher's exact test or χ2 test for categorical variables (α=0.05, two-tailed). Multivariable logistic regression models for dichotomous outcomes (adherence=no/yes) and multiple linear regression models for continuous outcomes (concentrations of/drugs in the hair) will be used to study the different factors associated with correct or non-adherence to therapy.

Multivariable analyses will aim to assess any correlation between adherence and clinical/demographic variables in an expository manner. Subsequently, it will be possible to evaluate in which classes of drugs there is a higher/lower adherence.

ELIGIBILITY:
Inclusion Criteria:

* All patients older than 18 years of both sexes with a diagnosis of hypertension undergoing treatment for at least 3 months with antihypertensive drugs and also statins.
* Diagnosis of secondary forms of hypertension excluded.
* Subjects who express their willingness to participate in the study by signing the consent form having understood the content of the written and verbal information provided about the purpose and mode of execution of the study.

Exclusion Criteria:

* Subjects unable to express voluntary adherence to the study.
* Renal insufficiency with estimated glomerular filtrate less than 50 mL/minute-
* Heart failure with functional class equal to or greater than II.
* Chronic inflammatory disease.
* Neoplastic disease.
* Any chronic diseases requiring continuous treatment with drugs known to interact pharmacokinetically with the antihypertensive drugs being monitored.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (n=200) followed for essential hypertension at the SIIA centres will be evaluated on the basis of their clinical characteristics, the presence of comorbidities and the therapeutic scheme in place and will be subjected to hair sampling for the analysis of drugs of interest and their possible metabolites in this matrix. The use of the prescribed drugs will be recorded along with the relevant clinical parameters and preliminarily evaluated by application of a questionnaire.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-05-15 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Determination of the concentration of antihypertensive drugs in hair samples collected at the first and second visits | 3 months
  Determination of drug concentration is used for the classification of patients as adherent or non-adherent to therapy or part of therapy based on the presence of quantifiable drugs in different segments of the hair sample representative of the time interval covered by the study
Determination of the concentration of statins prescribed to patient in hair samples collected at the first and second visits | 3 months
  In patients who have had a prescription of statins in addition to antihypertensive drugs, their quantification in hair samples will be used to define the adherence to therapy.

SECONDARY OUTCOMES:
Comparison the results of hair analysis performed at the first and second visits. | 3 months
  Comparison in adherence to therapy between hair analysis data performed at the first and second visits.
Comparison of adherence to therapy in the presence of change in therapy | 3 months
  Comparison of adherence to therapy in the presence of change in therapy with the evaluation of single compounds (both antihypertensives and statins) and comparison of adherence to therapy following the change from the use of single compounds or the same in polypill therapy (two or more active ingredients together) by comparison of hair analysis data performed at the first and second visits.
Analysis of the relationship between adherence to therapy and factors associated with the patient. | 3 months
  Analysis of the relationship between adherence to therapy and factors associated with the patient (age, demographic and anthropometric data, clinical conditions, prescription of other medications).
Assessment of the feasibility of hair analysis | 3 months
  Assessment of the feasibility of hair analysis involves comparison with data collected through questionnaires and a preliminary quantitative assessment of the analysis of prescribed medications in the hair.

CONTACTS AND LOCATIONS:
Overall Officials: Franco Tagliaro, MD, Principal Investigator — Univeristy of Verona
Locations (1):
- Azienda Ospedaliera Universitaria Integrata Verona, Verona, Italy

REFERENCES:
- [Result] UNODC, Vienna: Guidelines for Testing Drugs under International Control in Hair Sweat and Oral Fluid. https://www.unodc.org/documents/scientific/ST_NAR_30_Rev.3_Hair_Sweat_and_Oral_Fluid.pdf
- [Result] Bellows BK, Ruiz-Negron N, Bibbins-Domingo K, King JB, Pletcher MJ, Moran AE, Fontil V. Clinic-Based Strategies to Reach United States Million Hearts 2022 Blood Pressure Control Goals. Circ Cardiovasc Qual Outcomes. 2019 Jun;12(6):e005624. doi: 10.1161/CIRCOUTCOMES.118.005624. Epub 2019 Jun 5. PMID 31163981
- [Result] Naderi SH, Bestwick JP, Wald DS. Adherence to drugs that prevent cardiovascular disease: meta-analysis on 376,162 patients. Am J Med. 2012 Sep;125(9):882-7.e1. doi: 10.1016/j.amjmed.2011.12.013. Epub 2012 Jun 27. PMID 22748400
- [Result] Simpson SH, Eurich DT, Majumdar SR, Padwal RS, Tsuyuki RT, Varney J, Johnson JA. A meta-analysis of the association between adherence to drug therapy and mortality. BMJ. 2006 Jul 1;333(7557):15. doi: 10.1136/bmj.38875.675486.55. Epub 2006 Jun 21. PMID 16790458
- [Result] De Geest S, Sabate E. Adherence to long-term therapies: evidence for action. Eur J Cardiovasc Nurs. 2003 Dec;2(4):323. doi: 10.1016/S1474-5151(03)00091-4. No abstract available. PMID 14667488
- [Result] Haynes RB, McDonald H, Garg AX, Montague P. Interventions for helping patients to follow prescriptions for medications. Cochrane Database Syst Rev. 2002;(2):CD000011. doi: 10.1002/14651858.CD000011. PMID 12076376
- [Result] Mancia G, Rea F, Corrao G, Grassi G. Two-Drug Combinations as First-Step Antihypertensive Treatment. Circ Res. 2019 Mar 29;124(7):1113-1123. doi: 10.1161/CIRCRESAHA.118.313294. PMID 30920930
- [Result] OSMED L'uso dei farmaci in Italia Rapporto Nazionale Anno 2019 https://www.aifa.gov.it/-/rapporto-osmed-2019
- [Result] Weisser B, Predel HG, Gillessen A, Hacke C, Vor dem Esche J, Rippin G, Noetel A, Randerath O. Single Pill Regimen Leads to Better Adherence and Clinical Outcome in Daily Practice in Patients Suffering from Hypertension and/or Dyslipidemia: Results of a Meta-Analysis. High Blood Press Cardiovasc Prev. 2020 Apr;27(2):157-164. doi: 10.1007/s40292-020-00370-5. Epub 2020 Mar 26. PMID 32219670
- [Result] Williams B, Mancia G, Spiering W, Agabiti Rosei E, Azizi M, Burnier M, Clement DL, Coca A, de Simone G, Dominiczak A, Kahan T, Mahfoud F, Redon J, Ruilope L, Zanchetti A, Kerins M, Kjeldsen SE, Kreutz R, Laurent S, Lip GYH, McManus R, Narkiewicz K, Ruschitzka F, Schmieder RE, Shlyakhto E, Tsioufis C, Aboyans V, Desormais I; ESC Scientific Document Group. 2018 ESC/ESH Guidelines for the management of arterial hypertension. Eur Heart J. 2018 Sep 1;39(33):3021-3104. doi: 10.1093/eurheartj/ehy339. No abstract available. PMID 30165516
- [Result] Yusuf S, Joseph P, Dans A, Gao P, Teo K, Xavier D, Lopez-Jaramillo P, Yusoff K, Santoso A, Gamra H, Talukder S, Christou C, Girish P, Yeates K, Xavier F, Dagenais G, Rocha C, McCready T, Tyrwhitt J, Bosch J, Pais P; International Polycap Study 3 Investigators. Polypill with or without Aspirin in Persons without Cardiovascular Disease. N Engl J Med. 2021 Jan 21;384(3):216-228. doi: 10.1056/NEJMoa2028220. Epub 2020 Nov 13. PMID 33186492
- [Result] Scala D, Menditto E, Caruso G, Monetti VM, Orlando V, Guerriero F, Buonomo G, Caruso D, D'Avino M. Are you more concerned about or relieved by medicines? An explorative randomized study of the impact of telephone counseling by pharmacists on patients' beliefs regarding medicines and blood pressure control. Patient Educ Couns. 2018 Apr;101(4):679-686. doi: 10.1016/j.pec.2017.12.006. Epub 2017 Dec 9. PMID 29249596
- [Result] Raparelli V, Proietti M, Butta C, Di Giosia P, Sirico D, Gobbi P, Corrao S, Davi G, Vestri AR, Perticone F, Corazza GR, Violi F, Basili S. Medication prescription and adherence disparities in non valvular atrial fibrillation patients: an Italian portrait from the ARAPACIS study. Intern Emerg Med. 2014 Dec;9(8):861-70. doi: 10.1007/s11739-014-1096-1. Epub 2014 Jul 3. PMID 24990547
- [Result] Hassall D, Brealey N, Wright W, Hughes S, West A, Ravindranath R, Warren F, Daley-Yates P. Hair analysis to monitor adherence to prescribed chronic inhaler drug therapy in patients with asthma or COPD. Pulm Pharmacol Ther. 2018 Aug;51:59-64. doi: 10.1016/j.pupt.2018.07.001. Epub 2018 Jul 4. PMID 29981458
- [Result] Papaseit E, Marchei E, Mortali C, Aznar G, Garcia-Algar O, Farre M, Pacifici R, Pichini S. Development and validation of a liquid chromatography-tandem mass spectrometry assay for hair analysis of atomoxetine and its metabolites: Application in clinical practice. Forensic Sci Int. 2012 May 10;218(1-3):62-7. doi: 10.1016/j.forsciint.2011.10.012. Epub 2011 Oct 22. PMID 22024657
- [Result] Ferrari A, Licata M, Rustichelli C, Baraldi C, Vandelli D, Marchesi F, Palazzoli F, Verri P, Silingardi E. Monitoring of adherence to headache treatments by means of hair analysis. Eur J Clin Pharmacol. 2017 Feb;73(2):197-203. doi: 10.1007/s00228-016-2163-5. Epub 2016 Nov 20. PMID 27866243
- [Result] Gerona R, Wen A, Chin AT, Koss CA, Bacchetti P, Metcalfe J, Gandhi M. Quantifying Isoniazid Levels in Small Hair Samples: A Novel Method for Assessing Adherence during the Treatment of Latent and Active Tuberculosis. PLoS One. 2016 May 18;11(5):e0155887. doi: 10.1371/journal.pone.0155887. eCollection 2016. PMID 27191185